CLINICAL TRIAL: NCT05923164
Title: Reliability And Validity Study Of MAP-BC Evaluation Tool In Turkish Language To Detect Myofascial Adhesions Among Women Under Breast Cancer Treatment
Brief Title: Reliability And Validity Study Of "The Evaluation Tool For Myofascial Adhesions In Patients After Breast Cancer" In Turkish Language
Acronym: MAP-BC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 23/337
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; Upper Extremity Dysfunction; Tissue Adhesion
Keywords: Myofascial adhesions; Breast Cancer; POSAS; MAP-BC Evaluation Tool; myofascial dysfunction; validity and reliability study
MeSH Terms: conditions — Breast Neoplasms; Tissue Adhesions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Cancer Patients: Patients who had undergone breast cancer surgery, aged between 18-75 years-old
  Interventions: Diagnostic Test: MAP-BC (Myofascial Adhesions in Patients after Breast Cancer) Evaluation Tool; Diagnostic Test: Patient And Observer Scar Assessment Scale ( Observer Subscale)

INTERVENTIONS:
Diagnostic Test: MAP-BC (Myofascial Adhesions in Patients after Breast Cancer) Evaluation Tool — It's a tool to evaluate scar tissues that occured after breast cancer treatment. It quantitatively measures myofascial adhesions. The degree of adhesion is scored for each area at 3 different depth levels (skin, superficial, deep) as a 4-point scale (0: no adhesion - 3: severe adhesion). Axillary scar, breast/mastectomy scar, m. pectoralis region, frontal chest wall, lateral chest wall, axilla and inframammary fold are evaluated separately. Sum of the scores from three levels of each area gives the total score. The minimal total score is: 0 and the maximum total score is 63.
Diagnostic Test: Patient And Observer Scar Assessment Scale ( Observer Subscale) — This assesment tool consists of two different scales evaluated by the observer and the patient.The observer scale rates five variables, which include vascularity, pigmentation, thickness, relief, pliability and surface area, between 1-10 points (1:normal skin). The total score ranges from 5 to 50.

SUMMARY:
The aim of this observational study is to translate the MAP-BC Evaluation Tool into Turkish by adapting it to Turkish society and to conduct a validity and reliability study in women who have received breast cancer treatment.

The main questions it aims to answer are:

* Are the same researcher's MAP-BC Evaluation Tool results similar at intervals to detect myofascial adhesions in breast cancer patients in Turkish population?
* Are the different researchers' MAP-BC Evaluation Tool results similar to detect myofascial adhesions in breast cancer patients in Turkish population?
* After comparing the results of Turkish version of both The Patient and Observer Scar Assessment Scale Observer Subscale and MAP-BC Evaluation Tool, is there a sufficient correlation between them?

DETAILED DESCRIPTION:
Breast cancer is the most frequently diagnosed malignancy in all over the world. Breast and axillary surgery, radiotherapy, hormone therapy and chemotherapy treatments may cause upper extremity dysfunction and pain which negatively affect quality of life and daily living activities of breast cancer patients.

Lymphedema, severe pain, decreased range of motion of shoulder joint, axillary web syndrome, myofascial trigger points and myofascial adhesions are the leading causes affecting upper extremity function in patients with breast cancer.

Myofascial dysfunction presents as a problem characterized by trigger points, adhesions, and limitation of myofascial tissue and tissue gliding.

Muscle manipulation during surgery, scar tissue, soft tissue adhesions, adaptive posture development following surgery and radiotherapy induced fibrosis can cause myofascial adhesions. However, there is not sufficient research or tools for the evaluation of scar tissue and adhesions.

Detection, quantitative measurement and scoring of myofascial adhesions in upper extremity dysfunctions after breast cancer treatment are important for both developing target-oriented treatment plan and evaluation of treatment effectiveness (myofascial therapy, physical therapy modalities).

The Patient and Observer Scar Assessment Scale is an evaluation tool utilized to detect scar tissue and was shown for reliable and valid in patients who have undergone breast cancer surgery. Its reliability and validity study for Turkish population has been done earlier.

A new diagnostic method called MAP-BC (Myofascial Adhesions in Patients after Breast Cancer) has been developed to evaluate scar tissue after breast cancer treatments and to quantitatively measure myofascial adhesions. Its reliability and validity have been proven in various countries, however, it is yet to be tested in Turkey.

The aim of this observational study is to translate the MAP-BC evaluation tool into Turkish by adapting it to Turkish society and to conduct a validity and reliability study in women who have received breast cancer treatment.

Firstly, the original version of MAP-BC will be translated into Turkish and its semantic and conceptual equivalence will be checked. Later it will be finalized by the committee consisting of two translators and four expert physiatrists.

For intra-rater reliability, the same researcher will re-evaluate patients at 14-days intervals.

For inter-rater reliability, 2 different researchers will evaluate the first 15 patients by using the Patient and Observer Scar Assessment Scale and MAP-BC tools unaware of each other's results. If the outcome of the two researchers evaluation are found in agreement at a reliable rate, then the study will be continued by a single researcher.

The convergent validity of the Turkish version of MAP-BC will be assessed by comparing the results of Turkish version of both the Patient and Observer Scar Assessment Scale observer subscale (Patient and Observer Wound Assessment) and MAP-BC. Their correlation will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients aged between 18-75 years who had undergone breast surgery
* providing a written consent to participate in the study

Exclusion Criteria :

* Patients who do not agree to participate the study
* Patients with active skin disease/infection which limits physical examination (palpation)
* Patients with a secondary breast cancer and/or metastasis

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Gender
Study Population: Patients, aged between 18-75 years, who have undergone breast cancer surgery, visiting our oncological rehabilitation outpatient clinic between August 2023 and March 2024
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
MAP-BC Evaluation Tool | 11 months
  This tool was developed to evaluate scar tissues that occured after breast cancer treatments. It quantitatively measures myofascial adhesions. The degree of adhesion is scored for each area at 3 different depth levels (skin, superficial, deep) as a 4-point scale (0: no adhesion - 3: severe adhesion). Axillary scar, breast/mastectomy scar, m. pectoralis region, frontal chest wall, lateral chest wall, axilla and inframammary fold are evaluated separately. Sum of the scores from three levels of each area gives the total score. The maximum score is 63. In Breast cancer patients, the inter-rater reliability of the detection of myofascial adhesions by palpation has been reported good to excellent.
POSAS | 11 months
  This assesment tool consists of two different scales evaluated by the observer and the patient. Its validity and reliability have been proven for the detection of scar tissue in patients who have undergone breast cancer surgery. The observer scale rates five variables, which include vascularity, pigmentation, thickness, relief, pliability and surface area, between 1-10 points (1:normal skin). The total score ranges from 5 to 50. The Turkish version of POSAS, whose validity and reliability studies were conducted, will be used in our study.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz Bahar Özdemir, Principal Investigator
Locations (1):
- Sultan 2. Abdulhamid Han Training and Research Hospital, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Truong PT, Lee JC, Soer B, Gaul CA, Olivotto IA. Reliability and validity testing of the Patient and Observer Scar Assessment Scale in evaluating linear scars after breast cancer surgery. Plast Reconstr Surg. 2007 Feb;119(2):487-94. doi: 10.1097/01.prs.0000252949.77525.bc. PMID 17230080
- [Background] Lewit K, Olsanska S. Clinical importance of active scars: abnormal scars as a cause of myofascial pain. J Manipulative Physiol Ther. 2004 Jul-Aug;27(6):399-402. doi: 10.1016/j.jmpt.2004.05.004. PMID 15319762
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] De Groef A, Van der Gucht E, Dams L, Evenepoel M, Teppers L, Toppet-Hoegars J, De Baets L. The association between upper limb function and variables at the different domains of the international classification of functioning, disability and health in women after breast cancer surgery: a systematic review. Disabil Rehabil. 2022 Apr;44(8):1176-1189. doi: 10.1080/09638288.2020.1800835. Epub 2020 Aug 8. PMID 32772650
- [Background] Seyyah M, Yurdalan SU. Cultural adaptation and validation of Patient and Observer Scar Assessment Scale for Turkish use. Burns. 2018 Aug;44(5):1352-1356. doi: 10.1016/j.burns.2018.02.026. Epub 2018 Mar 24. PMID 29580666
- [Background] De Groef A, Van Kampen M, Vervloesem N, De Geyter S, Dieltjens E, Christiaens MR, Neven P, Geraerts I, Devoogdt N. An evaluation tool for myofascial adhesions in patients after breast cancer (MAP-BC evaluation tool): Development and interrater reliability. PLoS One. 2017 Jun 9;12(6):e0179116. doi: 10.1371/journal.pone.0179116. eCollection 2017. PMID 28598978